CLINICAL TRIAL: NCT05076084
Title: Evaluation of the Efficacy and Safety of Tacrolimus 0.1% Ophthalmic Solution in Children With Vernal Keratoconjunctivitis Resistant to Ciclosporin 2% Ophthalmic Solution: a Single-center Retrospective Cohort Study
Brief Title: Evaluation of the Efficacy and Safety of Tacrolimus Drops in Children With Vernal Keratoconjunctivitis
Acronym: KERAVER
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RGR_2021_21
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: Vernal keratoconjunctivitis; Tacrolimus
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 0 to 18 years followed for Vernal keratoconjunctivitis: Treated (or having been treated) with tacrolimus 0.1% ophthalmic solution previously treated with ciclosporin 2% ophthalmic solution with treatment failure.
  Interventions: Procedure: QUICK questionnaire and 6 additional questions; Other: Retrospective collection of clinical data from the patients' medical records

INTERVENTIONS:
Procedure: QUICK questionnaire and 6 additional questions — QUICK questionnaire and 6 additional questions
Other: Retrospective collection of clinical data from the patients' medical records — Retrospective collection of clinical data from the patients' medical records

SUMMARY:
Non-interventional single-center cohort study (Rothschild Foundation Hospital) of patients aged 0 to 18 years followed up in ophthalmology for KCV, treated with tacrolimus 0.1% eye drops previously treated with ciclosporin 2% with treatment failure.

1. Prospective collection of quality of life from the parents and/or, if possible, the children via the QUICK questionnaire and 6 additional questions
2. Retrospective collection of clinical data (secondary endpoints) from the patients' medical records, aiming to compare the period before the start of treatment and the period under treatment with TALYMUS

The objective of this study is to evaluate the response to TALYMUS® treatment in patients with Vernal keratoconjunctivitis who have failed ciclosporin 2% therapy, whether due to lack of efficacy, compliance difficulties or poor tolerance.

DETAILED DESCRIPTION:
Vernal keratoconjunctivitis (VKC) is a chronic inflammatory eye disease affecting children and adolescents. It is a disease of allergic origin which, if left untreated, can have a significant impact on quality of life, daily activities and learning. In some cases, sequelae of the disease or complications from the treatments used can lead to permanent vision impairment.

Symptoms of VKC include intense itching, tearing, mucous secretions, burning, foreign body sensation and severe photophobia. Clinical signs include conjunctival and corneal involvement -which may leave scarring opacities-and in the most severe stage, limbal insufficiency with definitive corneal conjunctivalization.

There is no consensus on the therapeutic strategy to adopt. Treatment is based on a combination of antihistamines and mast cell stabilizers, and in case of failure on corticosteroids. Cortico-resistant or cortico-dependent forms require treatment with local or general immunosuppressants, because of the long-term ocular complications of corticosteroids. These local immunosuppressants, belonging to the class of calcineurin inhibitors, have been used in ophthalmology for many years in hospital preparations of ciclosporin eye drops. More recently, commercial forms have appeared on the market: RESTASIS® (0.05% cyclosporine eye drops), IKERVIS® and VERKAZIA® (0.1% cyclosporine eye drops), CICLOGRAFT® (2% cyclosporine eye drops) and TALYMUS® (0.1% tacrolimus eye drops).

Although TALYMUS® has French marketing authorization for VKC, its place in the therapeutic strategy and its positioning in relation to the various cyclosporine eye drops is not clearly established. Series have reported similar efficacy of TALYMUS® and 0.05% and 2% cyclosporine in patients with KCV, at a lower dosage than those usually required for cyclosporine eye drops (2 drops per day for TALYMUS® versus 3 to 4 drops per day for cyclosporine). Given the difficulties of compliance in children, particularly in a school environment and in the context of a chronic pathology, the possibility of a less frequent administration represents a significant advantage. The simplicity of use and efficacy of TALYMUS® , as well as its safety profile, which is comparable to that of cyclosporine eye drops, have led some authors to recommend it as a first-line eye drop on a par with cyclosporine.

In addition, in numerous publications and in our experience, there are cases of failure of treatment with cyclosporine eye drops, which have even led some authors to recommend for many years only hospital preparations of cyclosporine at concentrations greater than or equal to 1%. It is therefore to be expected that cases of resistance to VERKAZIA® will appear.

One study reported the efficacy of a 0.1% tacrolimus hospital preparation in patients who had failed 1% cyclosporine therapy. However, the efficacy of TALYMUS® treatment in patients who have failed ciclosporin 2% therapy has not been reported to date.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in ophthalmology for vernal keratoconjunctivitis .
* Treated (or having been treated) with tacrolimus 0.1% ophthalmic solution previously treated with ciclosporin 2% ophthalmic solution with treatment failure.

Exclusion Criteria:

* Parental opposition

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with vernal keratoconjunctivitis, treated (or having been treated) with tacrolimus 0.1% ophthalmic solution previously treated with ciclosporin 2% ophthalmic solution with treatment failure.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Quality of life with TALYMUS® ophthalmic solution versus ciclosporin 2% ophthalmic solution | Day 1
  Score distribution of the QUICK questionnaire with TALYMUS® ophthalmic solution versus ciclosporin 2% ophthalmic solution in children with vernal keratoconjunctivitis treated with TALYMUS® ophthalmic solution due to ciclosporin 2% failure

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Rebecca, Principal Investigator — Hôpital Fondation A. de Rothschild; Gilles MARTIN, Study Chair — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschuld, Paris, France